CLINICAL TRIAL: NCT05913505
Title: A Randomized Controlled Trial of Heart Rate Variability Biofeedback Following Traumatic Brain Injury
Brief Title: Heart Rate Variability Biofeedback Following Traumatic Brain Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham Young University (Other)
Responsible Party: Principal Investigator, Leah Talbert, Principal Investigator, Brigham Young University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TBI_HRVB
Record Dates: First submitted 2023-04-02; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Twenty-five participants will complete the treatment condition in a pseudo-randomized order (determined by random number generator with constraints) such that half of the participants will be given the heart rate variability biofeedback active condition and half will be given the sham control condition. However, the participants in the sham control condition will be offered treatment with heart rate variability biofeedback after study completion. The heart rate variability biofeedback active condition is designed to increase heart rate oscillations (Osc+ condition) consistent with current best practices, while the sham control heart rate variability biofeedback condition is designed to decrease heart rate oscillations (Osc- condition).
Who Masked: Participant, Outcomes Assessor
Masking Description: Baseline measurements will be collected by undergraduate research assistants blinded to group conditions to reduce possible experimenter bias effects. Additionally, research assistants will be blinded to conditions for all testing sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSC+ (Experimental): Twenty-five participants will complete five weeks of heart rate variability biofeedback using emWave software (HeartMath®Institute, 2020). Participants will receive a weekly 30-minute heart rate variability biofeedback session for five weeks at the University Parkway Center, Brigham Young University. The heart rate variability biofeedback protocol will be based on Lehrer et al., 2013 and Yoo et al., 2022. This format will aid participants in implementing and learning breathing and heart rate variability biofeedback skills (Lehrer et al., 2020). All participants will wear an ear sensor to measure their pulse. The heart rate variability biofeedback will focus on autonomic balance through slow breathing at a resonance frequency of approximately 6 breathes per minute. The best approximate breathing pace for resonance frequency will be estimated and participant's resonance frequency will be provided and used for their homework and subsequent training sessions.
  Interventions: Behavioral: OSC+
- OSC- (Sham Comparator): Twenty-five participants will complete five weeks of Osc-. Similarly, for the Osc- procedures, the client will be required to complete a five-week intervention. During the weekly session, participants will also be wearing an earlobe monitor with HeartMath. Participants will be administered the Scale of Positive and Negative Experience at the beginning of each session to assess for mood. Participants will also be administered the 3-item Rivermead Post Concussion Symptoms Questionnaire at the beginning of each session. Participants will be instructed that the purpose of this portion of the study is to decrease their breathing oscillations. A program was designed by Yoo and colleagues (2022) that gives feedback regarding a "calmness" score which reflects a better score (i.e., higher) when participants breath in a pattern that elicits less variability (i.e., less oscillations).
  Interventions: Behavioral: OSC-

INTERVENTIONS:
Behavioral: OSC+ — The first session of the HRVB intervention will focus on introducing the client to HRVB and calculating the participant's resonance frequency which typically range from 4.5-7 breaths per minute. Participants will first complete a five-minute baseline breathing condition. Following the breathing condition, the participants will complete five conditions for five minutes each. Specifically, each condition will have the person breath at 6, 6.5, 5.5, 5, and 4.5 breaths per minute with a minute break between. Session two will focus on practicing resonance frequency breathing and solidifying the correct resonance frequency for the participant. Additionally, this session will introduce the technique of breathing through pursed lips and abdominal breathing. For sessions three through five, participants will practice resonance frequency breathing and review previous strategies.
  Arms: OSC+
Behavioral: OSC- — During the first week, the baseline will be assessed and resonance frequency. Specifically, during their first intervention session the participants will be told that the goal of the sessions includes decreasing heart rate variability and avoiding slow and steady breathing. The participants will then be asked to choose five strategies to lower their heart rate oscillations. Participants will be told to avoid slow breathing as it causes large heart rate oscillations. For the second session, the therapist will check in with the participant and discuss how the practice went. Participants will then select three strategies that they will practice for three five-minute conditions following a five-minute baseline. Sessions three, four, and five will include three conditions: a five-minute baseline and two strategies of their choice. For each session, the best strategy will be calculated and written on the assignment sheets to be used during the week for their four homework sessions.
  Arms: OSC-

SUMMARY:
Individuals with mild traumatic brain injury will be randomly assigned to an active heart rate variability biofeedback condition and a sham condition. The investigators will use a randomized pre-post design that will consist of two data collection phases and a 5-week treatment condition. The heart rate variability biofeedback active condition is designed to increase heart rate oscillations (Osc+ condition) consistent with current best practices, while the sham control heart rate variability biofeedback condition is designed to decrease heart rate oscillations (Osc- condition).

DETAILED DESCRIPTION:
There are two primary aims of the study: (1) examine whether heart rate variability increases at rest in individuals with mild traumatic brain injury from pre-treatment to post-treatment following heart rate variability biofeedback; (2) to test whether heart rate variability recovery following a stressor improves in individuals with mild traumatic brain injury following heart rate variability biofeedback. Regarding the first primary aim, the investigators hypothesize that heart rate variability will be higher in individuals with mild traumatic brain injury following heart rate variability biofeedback compared to those in the control/sham condition where the investigators do not expect such improvement pre- to post-testing. For the second aim, consistent with previous work, the investigators hypothesize that heart rate variability recovery following a stressor will be faster in individuals with mild traumatic brain injury following heart rate variability biofeedback compared to a sham control condition. There are three secondary aims for this study: (1) to evaluate whether improvements in heart rate variability in individuals with mild traumatic brain injury following heart rate variability biofeedback are associated with improvements in physical symptoms common after head injury (i.e., headaches, dizziness, sleep disturbance); (2) to evaluate whether improvements in heart rate variability in individuals with mild traumatic brain injury following heart rate variability biofeedback are associated with improvements in emotional functioning (i.e., life satisfaction, anxiety symptoms, depression symptoms); and (3) to evaluate whether improvements in heart rate variability in individuals with mild traumatic brain injury following heart rate variability biofeedback are associated with improvements in cognitive functioning (i.e., attention, inhibitory control).

ELIGIBILITY:
Inclusion Criteria:

* At least six months post-injury to account for spontaneous recovery
* Aged 18-55 years
* Fluent in English
* Able to provide informed consent.

Exclusion Criteria:

* Presence of a pacemaker
* Previous self-reported heart attack with hospitalization
* Diagnosed learning disability
* Other neurological difficulties or diagnoses (i.e., stroke, epilepsy)
* Participation in current litigation
* Uncorrected visual impairment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-04-24 (Estimated); Study Completion 2024-04-24 (Estimated)

PRIMARY OUTCOMES:
Stress Recovery | Through study completion, an average of 7 weeks
  Test whether heart rate variability recovery following a stressor improves in individuals with mild traumatic brain injury following heart rate variability biofeedback
Resting HRV | Through study completion, an average of 7 weeks
  Examine whether heart rate variability increases at rest in individuals with mild traumatic brain injury from pre-treatment to post-treatment following heart rate variability biofeedback

SECONDARY OUTCOMES:
Physical Symptoms | Through study completion, an average of 7 weeks
  The Rivermead Post Concussion Symptoms Questionnaire is a 16-item self-report measure of the severity of post-concussive symptoms following traumatic brain injury. The scale includes three categories of behavioral, physical, and cognitive symptoms, where participants are asked to rate the degree to which they experience 16 concussive symptoms in comparison to pre-injury symptoms within the past 24 hours. The items are rated on a 5-point scale from 0 (not experienced at all) to 4 (a severe problem). The RPQ-13 and RPQ-3 have good internal consistency and good test-retest reliability (0.89 and 0.72, respectively).
Scale of Positive and Negative Experience | Through study completion, an average of 7 weeks
  The Scale of Positive and Negative Experience is a 12-item scale that assesses participant experiences in various states (e.g., sad, happy, afraid) on a 5-point scale from 1 (never) to 5 (always).
Depression Anxiety Stress Scales | Through study completion, an average of 7 weeks
  The Depression Anxiety Stress Scales is a three-part self-report measure consisting of 42 items related to negative emotional states of tension/stress, anxiety, and depression. Each scale contains subscales of 2-4 items totaling 14 items. Each scale contains a four-point scale of severity and frequency to be rated on experiences over the past week.
Satisfaction with Life Scale | Through study completion, an average of 7 weeks
  The Satisfaction with Life Scale assesses judgments of one's life satisfaction using a 5-item scale. Scores are reported on a 7-point scale from 1 (strongly disagree) to 7 (strongly agree). While the scale does not assess life satisfaction across multiple domains, it quantifies a global measure of subjective well-being. Total scores range from 7 to 35, with higher scores indicating higher satisfaction.
Cognitive Functioning | Through study completion, an average of 7 weeks
  The NIH Toolbox for the Assessment of Neurological Behavior and Function Cognition Battery is approximately 30 minutes and consists of seven measures, including Picture Vocabulary, Oral Reading Recognition, Picture Sequence Memory, Dimensional Change Card Sort Test, List Sorting Working Memory, Flanker Inhibitory Control and Attention Test, and Pattern Comparison Processing Speed. The NIHTB-CB consists of two composite scores: a Crystallized Cognition Composite Score, providing a pre-injury estimate of overall cognitive ability, which is a combined score of Picture Vocabulary and Oral Reading Recognition; and a Fluid Cognition Composite Score, which is a combined score of Picture Sequence Memory, Dimensional Change Card Sort Test, List Sorting Working Memory, Flanker Inhibitory Control and Attention Test, and Pattern Comparison Processing Speed. The age-adjusted scaled score has a mean of 100 and a standard deviation of 15.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Larson, PhD, Study Chair — Brigham Young University
Locations (1):
- Brigham Young University, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, materials, and analysis plans are already posted on the Open Science Framework (https://osf.io/5gwpk). Actual study data (de-identified) will be made available, along with analysis codes, once the study has been complete and published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once data collection and data analysis has been completed and published in a scientific journal, the study data (de-identified) will either be posted on an open science website, such as the Open Science Framework, or will be given to other researchers upon request.
URL: http://osf.io/5gwpk